CLINICAL TRIAL: NCT03968367
Title: To Study the Effect of Magnetic Activated Sperm Sorting on the Outcome of in Vitro Fertilization-embryo Transplantation Among Patients With High DNA Fragmentation Index
Brief Title: To Study the Effect of Magnetic Activated Sperm Sorting on the Outcome of in Vitro Fertilization-embryo Transplantation
Acronym: MASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li-jun Ding (Other)
Responsible Party: Sponsor-Investigator, Li-jun Ding, Principal Investigator, Nanjing University
Organization: Nanjing University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-2018-MASS1
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Infertility, Male
Keywords: magnetic activated sperm sorting; DNA fragmentation index; sperm up; density differential centrifugation; clinical outcome
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic activated sperm cell sorting for infertile man (Experimental): A 0.5 mL aliquot of spermatozoa suspended in HTF-modified HEPES buffer, obtained either after sperm wash to remove the seminal plasma or after DGC, was centrifuged and the pellet (maximum of 107 cells) was resuspended in 80 uL of binding buffer with 20 uL of Annexin V-conjugated microspheres, both from the Annexin V microbead kit (Miltenyi Biotec, Huburn, CA, USA), for 15 min at room temperature. After addition of 400 lL of binding solution, the suspension was placed in the separation column (MiniMACS, Miltenyi Biotec). Labeled (apoptotic) cells were retained on the column and non-labeled (viable) cells passed through the column.
  Interventions: Procedure: Magnetic activated sperm sorting

INTERVENTIONS:
Procedure: Magnetic activated sperm sorting — MACS is a technique which allows the spermatozoa with the best characteristics to be selected for use in assisted reproduction treatments. This technique removes apoptotic spermatozoa - those which will die without achieving fertilisation - and selects the healthy ones, thus increasing the possibility of pregnancy.
  Other Names: Magnetic activated cell sorting

SUMMARY:
Recent studies have evaluated the use of magnetic-activated sperm sorting (MASS) to reduce apoptotic spermatozoa and improve the outcome of infertile male with assisted reproductive technology (ART). However, some results were inconsistent with above. The sperm of male with abnormal semen analysis tend to be accompanied with high apoptotic and high DNA fragmentation index (DFI). Hence, this study aimed at determining the efficiency of MASS in improving the clinical outcome of patients with high DFI).

DETAILED DESCRIPTION:
Patients will be recruited from our reproductive medicine center in Nanjing Drum towel Hospital, from July 2019 to July 2020. After semen analysis and selection of infertile men with at least two abnormal sperm parameters and obtaining the informed consent of the patients according to the admission criteria, the patients who enter the project will be randomly divided into the control group (n=30) whose sperm will be screened by density differential centrifugation (DGC) with swim up, and the observation group will be screened by MASS, followed by DGC. Then the procedure of in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) will be performed. Embryo transfer will be underwent according to the developmental speed and morphological characteristics of the embryo. The clinical outcomes after transplantation will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnostic as infertile according to 2007 WHO guidelines;
* DFI>25%.

Exclusion Criteria:

* With obvious female infertile factors;
* Sperm count <10 million;
* Chromosomal abnormalities in either or both of the couple;
* Loss of follow up or incomplete information of patients.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-19 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 2-3 months
  Pregnancy rate was defined from posi tive blood HCG and ultrasonography findings showing at least one embryo with a foetal heart beat 5 weeks after transfer.
Implantation rate | 2-3 months
  Implantation rate means the percentage of those embryos that implanted themselves into the uterine lining after having been transferred to the womb. Fetal heartbeat can be visualized via ultrasound in order to definitely confirm the implantation of the embryo.
Live-birth rate | 1year
  Live birth rate was defined as the number of deliveries that resulted in a live born neonate.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China